CLINICAL TRIAL: NCT06441487
Title: Evaluating a Remotely Delivered, Digital Health CRC Screening Intervention Among Racially Diverse Patients of a Community Health Center
Brief Title: mPATH-Cloud for Colorectal Cancer Screening
Acronym: mPATH-Cloud
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 23-1969; R01CA260822 (NIH)
Record Dates: First submitted 2024-05-22; First posted 2024-06-04 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer
Keywords: screening; digital health platform; mPATH™; Mobile Patient Technology for Health; fecal immunochemical tests; fecal occult blood test; Cancer Screening; Community Health Centers; Implementation Science; Rural health; Telemedicine; Minority Health
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized: Participants are assigned to intervention groups by chance.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial Mailed FIT Intervention (Experimental): Subjects randomized to this arm receive a link to a mobile health decision support tool (mPATH™-Cloud). Within mPATH™-Cloud, subjects are invited to answer brief questions to confirm eligibility, view a video to help them identify their CRC screening preference, and request either colonoscopy or fecal immunochemical test (FIT) screening from their primary care provider. Subjects who do not click on the link or select a screening test receive a FIT mailed to their home address.
  Interventions: Behavioral: Mobile Health Decision Support
- Trial Usual Care (Active Comparator): Subjects randomized to this arm receive usual care. Current usual care at the participating community health centers consists of a visit-based colorectal cancer screening recommendation and referral.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Mobile Health Decision Support — Subjects randomized to this arm receive a link to a mobile health decision support tool (mPATH™- Cloud). Within mPATH™-Cloud, subjects are invited to answer brief questions to confirm eligibility, view a video to help them identify their CRC screening preference, and request either colonoscopy or fecal immunochemical test (FIT) screening from their primary care provider. Subjects who select FIT, as well as subjects who do not click on the link or select a screening test receive a FIT mailed to their home address.
  Other Names: mPATH™-Cloud
  Arms: Trial Mailed FIT Intervention
Behavioral: Usual care — The study team will send subjects a prompt to visit the mobile health decision support tool (mPATH™-Cloud). Subjects with a mobile phone (as determined by their electronic health record) will receive a link to mPATH-Cloud by text. Subjects with a mailing address, but no mobile phone number in the EHR, will receive a letter inviting them to access mPATH-Cloud via URL code. Within mPATH-Cloud, subjects are invited to answer brief questions to confirm eligibility, view a video to help them identify their CRC screening preference, and request either colonoscopy or fecal immunochemical test (FIT) screening from their primary care provider. Subjects who do not click on the link or select a screening test receive a FIT.
  Arms: Trial Usual Care

SUMMARY:
This study assesses the effectiveness of colorectal cancer (CRC) screening intervention, mobile Patient Technology for Health (mPATH™-Cloud), compared to usual care among subjects who are overdue for CRC screening according to recommendations of the United States Preventive Services Taskforce (USPSTF). The trial randomly selects and enrolls 1,000 eligible subjects served by one federally qualified health center (FQHC) in North Carolina. Subjects are randomized to two study arms, Usual Care (Arm 1) or Mobile Health Decision Support (Arm 2).

Usual care consists of a visit-based screening recommendation to complete a stool test (e.g., FOBT, FIT, Cologuard) or referral to a screening colonoscopy. Subjects randomized to the Mobile Health Decision Support (Arm 2) are sent a message by text or US mail, depending on their preferred communication mode as indicated in the electronic health record (EHR), to visit the mPATH™-Cloud website. Subjects who engage with mPATH™-Cloud are invited to answer brief questions to confirm their eligibility and then view a short decision aid video designed to help people choose the CRC screening test (FIT or colonoscopy) that they would like to receive. After watching the video, subjects can choose a CRC screening test. Their primary care provider at the FQHC orders the appropriate test and, where indicated, refers the subjects to a colonoscopy. Subjects who request FIT screening and subjects who do not select any test receive a FIT mailed to their home address.

The primary outcome of interest is CRC screening completion within 6 months after randomization as assessed by EHR chart review. A completed screening is any of the following: colonoscopy completion (regardless of indication); 2) at least one FIT test with a normal result; or diagnostic colonoscopy following an abnormal FIT result. We hypothesize that we will observe a higher CRC screening completion rate in the Mobile Health Decision Support intervention arm (Arm 2).

This study includes up to three annual rounds of screening eligibility assessment and outreach. Repeated intervention rounds allow us to evaluate whether the intervention can improve adherence to USPSTF recommendations over time. During the 3-year intervention phase, Arm 1 receives usual care only.

DETAILED DESCRIPTION:
Subjects randomized to the Mobile Health Decision Support intervention arm (Arm 2) receive a link to mobile Patient Technology for Health (mPATH™-Cloud), a digital health platform designed to alleviate the implementation burden on clinical teams by automating many key steps in the CRC screening process. If the subject uses mPATH-Cloud to select a screening test, mPATH-Cloud notifies the subject's primary care provider at the FQHC. Subjects who request colonoscopy are then referred by their primary care provider to colonoscopy as appropriate. Subjects who request FIT receive a FIT mailed to their home.

Primary outcome assessment: To assess intervention effectiveness, CRC screening completion within 6 months of randomization (primary outcome) is assessed by EHR chart review. Screening completion is defined as any of the following: colonoscopy completion (regardless of indication); at least one FIT test with a normal FIT result; or diagnostic colonoscopy following an abnormal FIT result.

Secondary outcome assessment: To assess intervention effectiveness on adherence to USPSTF recommendations over time (secondary outcome), the Mobile Health Decision Support intervention is offered annually to Arm 2 subjects for up to 3 consecutive years so long as the subject remains eligible and due for CRC screening as determined by EHR review.

CRC screening up-to-datedness will be assessed by EHR chart review over a period of three consecutive years. FIT should be repeated annually, and colonoscopy typically only needs to be repeated once every 10 years. Thus, subjects will be assigned one year per annual FIT completed (e.g., FIT in years 1, 2, and 3 would be assigned 3 years; FIT in year 1, and 3 would be assigned 2 years) and up to 3 years for colonoscopy depending on the year received (e.g., colonoscopy in year 1 would be assigned 3 years, colonoscopy in year 3 would be assigned 1 year). Subjects remain in their originally assigned study arms for the duration of up to three annual rounds of CRC screening outreach.

Implementation assessment (exploratory outcome): This study will identify implementation processes and outcomes that will impact future dissemination and scalability. After the trial phase concludes, researchers will interview a subsample of up to 50 subjects to understand factors associated with CRC screening completion among subjects with varying needs and preferences.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-73 years at time of enrollment
* At average risk for CRC ("average risk" is defined as those subjects who do not have any of the following: documented history in the EHR of CRC, colonic adenomas, family history of CRC, or diagnosis of inflammatory bowel disease)
* No record in the EHR of fecal occult blood test (FOBT)/FIT within 12 months, FIT-DNA within 3 years, colonoscopy within 10 years, sigmoidoscopy within 5 years, barium enema within 5 years, or computed tomography (CT) colonography within 10 years of the EHR query date
* No record in the EHR of any CRC diagnosis or total colectomy
* Active patient of the clinic as documented in the EHR (seen at least 2 times within the past 12 months)
* For the second and third study rounds only: No record of a positive (abnormal) CRC screening result in a previous study round

Exclusion Criteria:

* All individuals meeting any of the exclusion criteria at baseline will be excluded from study participation:
* Age younger than 45 years or older than 73 years at the time of enrollment
* Not at average risk for CRC ("average risk" is defined as those subjects who do not have any of the following: history with colorectal carcinoma, colonic adenomas, family history of colorectal carcinoma, or diagnosis of inflammatory bowel disease)
* Colorectal carcinoma screening in last 12 months Record in the electronic health record (HER) of fecal occult blood test (FOBT)/FIT within 12 months, FIT-DNA within 3 years, colonoscopy within 10 years, sigmoidoscopy within 5 years, barium enema within 5 years, or computed tomography (CT) colonography within 10 years of the EHR query date
* Record in the EHR any CRC diagnosis or total colectomy
* Not an active client of the clinic as documented in the EHR (not seen at least 2 times within the past 12 months)
* For second and third annual study rounds only: Record of a positive (abnormal) CRC screening result in a previous study round

Ages: 45 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Colorectal cancer screening completion rate | Up to 6 months
  The proportion of individuals who completed CRC screening using any of the screening modalities recommended by the United States Preventive Service Task Force. Screening modalities could be fecal occult blood test (FIT), fecal occult blood test (FOBT), the stool DNA test combines the FIT ( FIT-DNA), colonoscopy, flexible sigmoidoscopy, flexible sigmoidoscopy with FIT, Computerized Tomography (CT) colonography.

SECONDARY OUTCOMES:
Colorectal cancer screening up-to-datedness | Baseline,1 year, 2 years, 3 years
  Colorectal cancer screening coverage at the time of annual assessment. screening modalities recommended by the United States Preventive Service Task Force. Screening modalities could be fecal occult blood test (FIT), fecal occult blood test (FOBT), the stool DNA test combines the FIT ( FIT-DNA), colonoscopy, flexible sigmoidoscopy, flexible sigmoidoscopy with FIT, Computerized Tomography (CT) colonography.

CONTACTS AND LOCATIONS:
Overall Officials: Leah M Frerichs, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Lineberger Comphrehensive Cancer Center at University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No
All of the participant data collected during the trial, after de-identification, will be made available.
  IPD Sharing Supporting Information Type: Study Protocol, SAP, and Analytic Code.
  IPD Sharing Time Frame: Beginning 6 months after summary data are published or otherwise made available with no end date.
  IPD Sharing Access Criteria: Investigators who provide a methodologically sound proposal to achieve aims in the approved proposal. Proposals should be directed to leahf@unc.edu.

REFERENCES:
- [Derived] Frerichs L, Zhang Z, Moore AA, Falk I, Tan X, Randazzo A, Brenner AT, S Reuland D, Dharod A, Miller DP Jr. Using a digital health platform to implement a multi-component CRC screening intervention within a federally qualified health center: study protocol for a hybrid type I trial. BMC Health Serv Res. 2025 Aug 8;25(1):1047. doi: 10.1186/s12913-025-13262-y. PMID 40781671
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials